CLINICAL TRIAL: NCT07067814
Title: The Identification of Recurrent Laryngeal Nerve by Injection of Methylene Blue Dye Into the Inferior Thyroid Artery in Comparison to The Conventional Technique During Thyroidectomy, Comparative Study
Brief Title: Comparison Between Two Techniques During Thyroidectomy (Conventional Dissection Technique and Injection of Methylene Blue Dye Into Inferior Thyroid Artery Technique) Regarding Recurrent Laryngeal Nerve Identification and Preservation
Acronym: RLN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD17/2023
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-05

CONDITIONS: Time Taken for Identification of Single Recurrent Laryngeal Nerve; Intra-operative Blood Loss
Keywords: Recurrent laryngeal nerve identification

STUDY DESIGN:
Intervention Model Description: 1. : - Methylene blue group: After ligation of the superior thyroid pole, 0.5-1 ml of sterile methylene blue dye was injected into the inferior thyroid artery. The thyroid tissue absorbed the dye, while the RLN remained unstained, appearing as a white structure in the tracheoesophageal groove. This aided in its early and safe identification, reducing the risk of injury during dissection.
  2. : Conventional technique group: the RLN was identified based on conventional anatomical landmarks without the use of dye. The nerve was traced along its expected course near the inferior thyroid artery and ligament of Berry
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylene blue group (Active Comparator): After ligation of the superior pole, 0.5-1 ml of sterile methylene blue dye was injected into the inferior thyroid artery. The thyroid tissue absorbed the dye, while the RLN remained unstained, appearing as a white structure in the tracheoesophageal groove. This aided in its early and safe identification, reducing the risk of injury during dissection.
  Interventions: Drug: Methylene blue group; Procedure: Methylene blue group
- Conventional technique group (No Intervention): the RLN was identified based on conventional anatomical landmarks without the use of dye. The nerve was traced along its expected course near the inferior thyroid artery and ligament of Berry

INTERVENTIONS:
Drug: Methylene blue group — After ligation of the superior pole, 0.5-1 ml of sterile methylene blue dye was injected into the inferior thyroid artery. The thyroid tissue absorbed the dye, while the RLN remained unstained, appearing as a white structure in the tracheoesophageal groove. This aided in its early and safe identification, reducing the risk of injury during dissection.
  Arms: Methylene blue group
Procedure: Methylene blue group — After ligation of the superior pole, 0.5-1 ml of sterile methylene blue dye was injected into the inferior thyroid artery. The thyroid tissue absorbed the dye, while the RLN remained unstained, appearing as a white structure in the tracheoesophageal groove. This aided in its early and safe identification, reducing the risk of injury during dissection.
  Arms: Methylene blue group

SUMMARY:
The aim of the study is to evaluate the value of injection of methylene blue dye into the inferior thyroid artery for the help of the identification and dissection of recurrent laryngeal nerve, so thyroidectomy could be done with fewer complications in comparison to conventional technique

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effectiveness of methylene blue dye injection into the inferior thyroid artery for enhancing the intraoperative visualization of the RLN during thyroidectomy. Also, this method was compared to conventional RLN identification techniques in terms of nerve identification time, blood loss, complication rates, and postoperative outcomes, while assessing the safety and feasibility of using methylene blue in thyroid surgery.

The study included 40 patients with indications for thyroidectomy due to benign thyroid conditions. Patients were randomly assigned into two equal groups:

* Group A: 20 patients underwent injection of methylene blue dye into the inferior thyroid artery to aid in identifying the recurrent laryngeal nerve (RLN).
* Group B: 20 patients underwent conventional RLN identification during thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* All patients who present with simple nodular goiter, solitary thyroid nodule, controlled toxic goiter and failed medical treatment with indication for thyroidectomy.
* Patents undergoing primary surgery (not recurrent).
* Patients who are willing to undergo surgery under general anesthesia without any preoperative complications or major diseases.
* Either gender in the age group of 18-60 years

Exclusion Criteria:

* Previous thyroid surgery.
* Malignant goiter.
* Major cardiac diseases, renal diseases or patients who are unfit for surgery.
* Methylene blue allergies.
* Pregnancy.
* Patients who refuse to participate in the study.
* Presence of any preoperative cord pathology or patients with dysphonia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Easy and fast identification of recurrent laryngeal nerve | Procedure (Time taken for identification of the recurrent laryngeal nerve after delivery of thyroid lobe (in minutes))
  Thyroid gland absorbed the dye and got stained blue while the RLN didn't take the dye and appeared as a white structure in the tracheoesophageal groove

SECONDARY OUTCOMES:
Lower intra-operative blood loss | The duration of the procedure ranging from one to two hours
  Intra-operative blood loss was significantly lower in the Methylene blue group in comparison to conventional technique

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet